CLINICAL TRIAL: NCT02633163
Title: A Phase II Controlled Trial of Allogeneic Mesenchymal Stem Cells for the Treatment of Refractory Lupus
Brief Title: Phase 2 Trial of Mesenchymal Stem Cells in Systemic Lupus Erythematosus (MiSLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUSC-UCMSC-001
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Stem Cell; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Mesenchymal Stem Cells (MSCs) (Experimental): Mesenchymal Stem Cells (MSCs) 1 x 10^6 cells/kg in Plasma-Lyte A solution
  Interventions: Drug: Low Dose Mesenchymal Stem Cells (MSCs)
- High Dose Mesenchymal Stem Cells (MSCs) (Experimental): Mesenchymal Stem Cells MSCs 5 x 10^6 cells/kg in Plasma-Lyte A solution
  Interventions: Drug: High Dose Mesenchymal Stem Cells (MSCs)
- Plasma Lyte A Solution (Placebo Comparator): Placebo Infusion (Plasma-Lyte A solution only)
  Interventions: Drug: Placebo Infusion

INTERVENTIONS:
Drug: Low Dose Mesenchymal Stem Cells (MSCs) — Participants will receive a single IV infusion of Mesenchymal Stem Cells (MSCs) 1 x 10^6 cells/kg in Plasma-Lyte A solution. All participants will receive the infusion at the Baseline (Day 0) visit. All participants will continue on their standard-of-care therapy during the trial.
  Arms: Low Dose Mesenchymal Stem Cells (MSCs)
Drug: High Dose Mesenchymal Stem Cells (MSCs) — Participants will receive a single IV infusion of Mesenchymal Stem Cells MSCs 5 x 10^6 cells/kg in Plasma-Lyte A solution.
  Arms: High Dose Mesenchymal Stem Cells (MSCs)
Drug: Placebo Infusion — Participants will receive a placebo infusion that does not contain any mesenchymal stem cells.The placebo infusion will consist of Plasma-Lyte A, which is the same vehicle used to deliver the MSCs in the experimental groups.
  Arms: Plasma Lyte A Solution

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mesenchymal stem cells (MSCs) obtained from umbilical cords for the treatment of adults with systemic lupus erythematosus (SLE). The goal of this study is to determine if patients receiving an MSC infusion plus standard of care respond better than patients receiving placebo infusion plus standard of care.

DETAILED DESCRIPTION:
A phase 2 multicenter (several medical research centers participating), placebo controlled, randomized (assigned by chance), double blind (neither the participant nor the investigator will know if active drug or placebo is assigned) trial to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) for the treatment of systemic lupus erythematosus (SLE) in adults.

The MSCs will be obtained from healthy donor umbilical cords and two doses of MSCs will be tested. The cells will be produced at the Medical University of South Carolina (MUSC) and will be shipped to other participating centers for patients with SLE. Participants will receive either active drug or placebo through a single IV infusion. All participants will receive standard of care and their safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old, male or female, of any race
* Historical presence of at least 4 of 11 of the ACR Classification Criteria
* Evidence of a positive ANA (≥1:80 titer) or positive dsDNA antibody test within 6 months of screening
* Clinically active SLE determined by SLEDAI score ≥6 and the presence of at least one BILAG A or BILAG B at screening, despite standard-of-care therapy
* If the patient has a BILAG A or BILAG B score in the renal organ system, he/she must have completed at least 6 months of therapy for the current episode of nephritis prior to Screening. Therapy must include at least 6 months of mycophenolate or at least 3 months of cyclophosphamide followed by mycophenolate or azathioprine
* Able and willing to give written informed consent

Exclusion Criteria:

* Active CNS lupus affecting mental status
* Active lupus nephritis requiring dialysis
* Laboratory exclusions: eGFR <30, WBC <2.0/mm3, hemoglobin <8 g/dL, platelet count <30,000/mm3, liver enzymes AST or ALT >4 times upper limit normal.
* Positive testing for HIV, hepatitis B or hepatitis C, tuberculosis (TB), or chest X-ray (CXR) findings consistent with TB or latent fungal infection.
* History of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix
* Pregnant or breast feeding
* A woman of childbearing potential (not post-menopausal or surgically sterile) who is not willing to use adequate contraception
* History of renal transplantation
* Herpes zoster within the past 90 days or any infection requiring hospitalization or intravenous or intramuscular antibiotics within the past 60 days
* Clinically significant EKG or chest X-ray changes
* Any other medical condition, related or unrelated to SLE, that in the opinion of the investigator would render the patient inappropriate or too unstable to complete study protocol
* Use of prednisone >0.5 mg/kg/day (or equivalent corticosteroid) within 1 month of Baseline visit
* Change or addition to immunosuppressant regimen within 3 months of Baseline visit (except corticosteroids); Use of other experimental therapeutic agents within 3 months of Baseline visit
* Having received belimumab within 2 months of Baseline, or having received rituximab or other B cell depleting biologic therapy within 6 months of Baseline.
* Comorbidities requiring corticosteroid therapy
* Current substance abuse or recent (within one year) history of substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2026-02-03 (Actual)

PRIMARY OUTCOMES:
Clinical response at Week 24 as defined by the SLE Responder Index (SRI): | Week 24
  Systemic Lupus Erythematosus Responder Index (SRI) is defined as a greater than or equal to (≥) 4 point reduction in the Systemic Lupus Erythematosus Disease Activity Index score (SLEDAI), no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B domain score, and no deterioration from Baseline in the Physician's Global Assessment (PGA) by greater than or equal to (≥) 0.3 points.
  Additionally, to be a "responder", corticosteroid dose must be less than of equal to (≤)10 mg/day of prednisone or equivalent by the Week 20 visit and be maintained at less than or equal to 10 mg/day through Week 24.

SECONDARY OUTCOMES:
Change in SLEDAI score between groups | Baseline to Weeks 12, 24, and 52
  Changes in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) between the experimental and placebo group.
Renal and non-renal organ system flares | At or before Weeks 12, 24, and 52
  Frequency of renal and non-renal organ system flares at or before Weeks 12, 24, and 52, defined by the BILAG criteria.
Changes in SLICC-DI | Baseline to Week 52
  • Change in SLICC-DI from Baseline to Week 52 to assess for accumulation of new damage (SLE-related or treatment-related)
Changes in HR-QOL | Baseline to Week 52
  Changes in HR-QOL (measured by SF36 v2) from Baseline to Weeks 12, 24, and 52
Changes in Fatigue | Baseline to Week 52
  Changes in fatigue (measured by PROMIS Fatigue Short Form (SF)) from Baseline to Weeks 12, 24, and 52
Changes in Pain | Baseline to Week 52
  Changes in pain (measured by PROMIS Pain SF) from Baseline to Weeks 12, 24, and 52
Changes in Depression | Baseline to Week 52
  Changes in depression (measured by PROMIS Depression SF) from Baseline to Weeks 12, 24, and 52
Changes in patient-reported lupus-specific disease status | Baseline to Week 52
  Changes in patient-reported lupus-specific disease status (measured by the LupusPro and LIT) from Baseline to Weeks 12, 24, and 52
Steroid-sparing effect | Baseline to Week 52
  Steroid-sparing effect (measured by discontinuation of corticosteroids and time to discontinuation among those taking corticosteroids)
Cumulative systemic steroid dose | Week 52
  Cumulative systemic steroid dose (PO, IV, IM) at Week 52
Changes in the presence of serum and urine biomarkers of SLE activity: | Baseline to Week 52
  Changes in the presence of serum and urine biomarkers of SLE activity: SLE-related cytopenias, low serum complement levels, anti-dsDNA levels or urine protein measures from Baseline to Weeks 12, 24, and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Gary S. Gilkeson, MD, Principal Investigator — Medical University of South Carolina; Diane L. Kamen, MD, MSCR, Study Chair — Medical University of South Carolina
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - San Diego, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina